CLINICAL TRIAL: NCT00801944
Title: Solifenacin in the Treatment of Urgency Symptoms of Overactive Bladder in a Rising Dose, Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Solifenacin Succinate 5mg or 10mg Once Daily in the Treatment of Urgency Symptoms
Acronym: SUNRISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 905-EC-002
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Solifenacin succinate 5/10mg
  Interventions: Drug: Solifenacin succinate
- II (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solifenacin succinate — oral
  Other Names: YM905; Vesicare
  Arms: I
Drug: Placebo — oral
  Arms: II

SUMMARY:
Prospective, double-blind, double-randomised, 2-arm parallel group study. Optimal dose increase. Primary efficacy assessment of OAB symptoms by patient diaries.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to complete the micturition diary correctly.
* Symptoms of overactive bladder (including urinary frequency, urgency with/without urge incontinence) for >= 3 months
* At least 3 episodes of urgency with or without incontinence in last 3 days
* At least three episodes of urgency with or without incontinence (PPIUS grade 3 or 4) during the 3-day micturition diary period
* Patient must experience frequency of micturition on average >= 8 times per 24-hour period during the 3-day micturition diary period

Exclusion Criteria:

* Pregnant women or women who intend to become pregnant during the study or women of childbearing potential who are sexually active and practising an unreliable method of birth control or will be lactating during the study. Reliable contraceptive methods are intra-uterine devices, contraceptive pills of combination type, hormonal implants and injectable or patch contraceptives
* Clinically significant outflow obstruction (at the discretion of the investigator)
* Significant post void residual volume (PVR>200ml)
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the investigator
* Patient with indwelling catheters or practising intermittent self-catheterisation
* Evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Hypersensitivity to solifenacin or to any of the excipients, uncontrolled narrow angle glaucoma, myasthenia gravis, urinary or gastric retention, severe renal impairment (GFR ≥30 ml/min), moderate or severe hepatic impairment, chronic intestinal disease, megacolon, requirement for dialysis, concomitant use of a strong CYP3A4 inhibitor, e.g. ketoconazole
* Non drug OAB treatment such as bladder-training, biofeedback and pelvic floor exercises are permissible if established at least 4 weeks prior to study start and intended to be continued throughout the study; electrostimulation therapy is not permissible at any time
* Use of drugs intended to treat urinary incontinence
* Diabetic neuropathy
* Any clinically significant condition, which in the opinion of the investigator makes the patient unsuitable for the trial
* Participation in any clinical trial within 30 days prior to randomisation
* Employees of the Yamanouchi Group, third parties associated with the study, or the study site
* Patient who did not complete the micturition diary according to the instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2004-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of urgency episodes/24 hours at EOS -from the Patient Perception of Intensity of Urgency Scale at void (PPIUS) grades 3 and 4 | Week 16

SECONDARY OUTCOMES:
Change from baseline in mean number of urgency episodes (PPIUS grades 1-4) | Week 16
Change from baseline in the mean number of micturition, incontinence and urge incontinence (PPIUS grade 4) episodes per 24 hours | Week 16
Change from baseline in patient perception of bladder condition (PBC) | Week 16
Change from baseline in patient perception of urgency 'bother' (UB-VAS) | Week 16
Percentage of patients requiring an increase in the dose of the study medication | Week 8
Patient assessment of treatment satisfaction (TS-VAS) | Weeks 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (78):
- Belgium (8):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Hasselt
  - Kortrijk
  - Leuven
  - Liège
- Czechia (3):
  - Ostrava
  - Prague
  - Zlín
- Al Mansurah, Egypt
- France (6):
  - Lille
  - Lomme
  - Mulhouse
  - Nantes
  - Nîmes
  - Paris
- Germany (14):
  - Aichach
  - Bad Neuenaher
  - Bamberg
  - Bautzen
  - Berlin
  - Dierdorf
  - Dülmen
  - Düsseldorf
  - Frankfurt
  - Henningsdorf
  - Munich
  - Neustadt
  - Nuremberg
  - Planegg
- Greece (3):
  - Athens
  - Crete
  - Ioannina
- Hungary (5):
  - Budapest
  - Nyíregyháza
  - Pécs
  - Szeged
  - Tatabánya
- Italy (8):
  - Bari
  - Catanzaro
  - Cinisello Balsamo
  - Magenta
  - Modena
  - Perugia
  - Turin
  - Udine
- Poland (2):
  - Bydgoszcz
  - Wroclaw
- Portugal (4):
  - Abrantes
  - Lisbon
  - Porto
  - Santarém
- Moscow, Russia
- Slovakia (3):
  - Banska Bysterica
  - Martin
  - Žilina
- Spain (7):
  - Barcelona
  - Coaña
  - Córdoba
  - Madrid
  - Mérida
  - San Cristóbal de La Laguna
  - Seville
- United Kingdom (13):
  - Birmingham
  - Cottingham
  - Croydon
  - Edinburgh
  - Huntingdon
  - London
  - Manchester
  - Oldham
  - Stoke-on-Trent
  - Sunderland
  - Torbay
  - Welwyn Garden City
  - Worthing

REFERENCES:
- [Background] Cardozo L, Hessdorfer E, Milani R, Arano P, Dewilde L, Slack M, Drogendijk T, Wright M, Bolodeoku J; SUNRISE Study Group. Solifenacin in the treatment of urgency and other symptoms of overactive bladder: results from a randomized, double-blind, placebo-controlled, rising-dose trial. BJU Int. 2008 Nov;102(9):1120-7. doi: 10.1111/j.1464-410X.2008.07939.x. Epub 2008 Oct 6. PMID 18990175
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401